CLINICAL TRIAL: NCT01095978
Title: Evaluation of the Treatment With Klacid SR in Patients With Acute Tracheitis, Tracheobronchitis and Bronchitis, Acute Exacerbation of Chronic Bronchitis and Mild Community-acquired Pneumonia in Common Clinical Practice in Ukraine
Acronym: KLARAINE
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Irina Magdik, Medical Director, Abbott Laboratories S.A., Ukraine
Other Study IDs: P11-979
Record Dates: First submitted 2010-02-28; First posted 2010-03-30 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Respiratory Tract Infections
Keywords: Klacid SR; Clarithromycin; Respiratory tract infections; Bronchitis; Pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis; Pneumonia | interventions — Clarithromycin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute upper respiratory tract diseases, bronchitis, pneumonia
  Interventions: Drug: Clarithromycin (Klacid SR)

INTERVENTIONS:
Drug: Clarithromycin (Klacid SR) — Klacid SR in a dose of 1000 mg once daily
  Other Names: Biaxin; Abbotic; Biclar; Klacid; Klaricid; Zeclar; Clarithromycin; Klacid SR

SUMMARY:
To describe the relief of symptoms, tolerability, and compliance of treatment with Klacid® sustained release (SR) at a dose of 1000 mg once daily in patients with acute tracheitis, acute tracheobronchitis, acute bronchitis, or in patients with acute exacerbation of chronic bronchitis or mild community-acquired pneumonia.

This postmarketing observational study is non-interventional and is being conducted in a prospective, single-arm, single-country, multicenter format.

Klacid SR will be prescribed in usual manner in accordance with the terms of the local market authorization with regards to dose, population, and indication as well as with local guidelines.

DETAILED DESCRIPTION:
The postmarketing observational study is observational in nature. Its follow-up is not interventional and is left to the judgment of each physician during the observational period, which defines the survey for each patient. Follow-up of patients should enable two patient visits during this period.

The screening/inclusion visit (Visit 1) will be performed when the decision for Klacid SR therapy in a daily dose of 1000 mg is made. The second visit of the patient will occur 10 - 16 days from the screening/inclusion Visit (upon physician's decision). The physician can change the numbers and time of the visits. As a result, failure to meet these suggested dates will not constitute a breach of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men, women 18 years with

  1. Acute tracheitis.
  2. Acute tracheobronchitis.
  3. Acute bronchitis.
  4. Mild community-acquired pneumonia.
  5. Acute exacerbation of chronic bronchitis.
* To whom decision to initiate Klacid SR therapy in a dose of 1000 mg has been made by physician.

Exclusion Criteria:

* Known hypersensitivity to macrolide antibiotics
* Documented renal impairment (creatinine clearance under 30 ml/min)
* Concomitant therapy with the following drugs: astemizole, cisapride, pimozide, terfenadine and ergotamine or dihydroergotamine
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consulting rooms of general practitioners, pulmonologists, and allergologists and centers with experience in the treatment of patients with acute upper respiratory tract diseases, acute bronchitis or acute exacerbation of chronic bronchitis or mild community-acquired pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 2822 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Magdik, MD, Study Director — Abbott Laboratories S.A., Ukraine
Locations (126):
- Ukraine (126):
  - Site Reference ID/Investigator# 29842, Dnipro
  - Site Reference ID/Investigator# 29848, Dnipro
  - Site Reference ID/Investigator# 30028, Dnipro
  - Site Reference ID/Investigator# 30046, Dnipro
  - Site Reference ID/Investigator# 30047, Dnipro
  - Site Reference ID/Investigator# 30049, Dnipro
  - Site Reference ID/Investigator# 30059, Dnipro
  - Site Reference ID/Investigator# 30074, Dnipro
  - Site Reference ID/Investigator# 30080, Dnipro
  - Site Reference ID/Investigator# 30099, Dnipro
  - Site Reference ID/Investigator# 30535, Dnipro
  - Site Reference ID/Investigator# 30572, Dnipro
  - Site Reference ID/Investigator# 30574, Dnipro
  - Site Reference ID/Investigator# 30575, Dnipro
  - Site Reference ID/Investigator# 30576, Dnipro
  - Site Reference ID/Investigator# 30577, Dnipro
  - Site Reference ID/Investigator# 30578, Dnipro
  - Site Reference ID/Investigator# 30579, Dnipro
  - Site Reference ID/Investigator# 30580, Dnipro
  - Site Reference ID/Investigator# 30581, Dnipro
  - Site Reference ID/Investigator# 30582, Dnipro
  - Site Reference ID/Investigator# 30583, Dnipro
  - Site Reference ID/Investigator# 30589, Dnipro
  - Site Reference ID/Investigator# 30590, Dnipro
  - Site Reference ID/Investigator# 30622, Dnipro
  - Site Reference ID/Investigator# 30623, Dnipro
  - Site Reference ID/Investigator# 30050, Donetsk
  - Site Reference ID/Investigator# 30051, Donetsk
  - Site Reference ID/Investigator# 30054, Donetsk
  - Site Reference ID/Investigator# 30057, Donetsk
  - Site Reference ID/Investigator# 30060, Donetsk
  - Site Reference ID/Investigator# 30066, Donetsk
  - Site Reference ID/Investigator# 30071, Donetsk
  - Site Reference ID/Investigator# 30073, Donetsk
  - Site Reference ID/Investigator# 30573, Donetsk
  - Site Reference ID/Investigator# 30584, Donetsk
  - Site Reference ID/Investigator# 30585, Donetsk
  - Site Reference ID/Investigator# 30600, Donetsk
  - Site Reference ID/Investigator# 30601, Donetsk
  - Site Reference ID/Investigator# 30586, Donetsk
  - Site Reference ID/Investigator# 30587, Donetsk
  - Site Reference ID/Investigator# 30588, Donetsk
  - Site Reference ID/Investigator# 29840, Kharkiv
  - Site Reference ID/Investigator# 30052, Kharkiv
  - Site Reference ID/Investigator# 30056, Kharkiv
  - Site Reference ID/Investigator# 30058, Kharkiv
  - Site Reference ID/Investigator# 30065, Kharkiv
  - Site Reference ID/Investigator# 30067, Kharkiv
  - Site Reference ID/Investigator# 30075, Kharkiv
  - Site Reference ID/Investigator# 30076, Kharkiv
  - Site Reference ID/Investigator# 30078, Kharkiv
  - Site Reference ID/Investigator# 30079, Kharkiv
  - Site Reference ID/Investigator# 30096, Kharkiv
  - Site Reference ID/Investigator# 30102, Kharkiv
  - Site Reference ID/Investigator# 30616, Kharkiv
  - Site Reference ID/Investigator# 30617, Kharkiv
  - Site Reference ID/Investigator# 30624, Kharkiv
  - Site Reference ID/Investigator# 30625, Kharkiv
  - Site Reference ID/Investigator# 30626, Kharkiv
  - Site Reference ID/Investigator# 30627, Kharkiv
  - Site Reference ID/Investigator# 30628, Kharkiv
  - Site Reference ID/Investigator# 30632, Kharkiv
  - Site Reference ID/Investigator# 30633, Kharkiv
  - Site Reference ID/Investigator# 40761, Kharkiv
  - Site Reference ID/Investigator# 30027, Kiev
  - Site Reference ID/Investigator# 30097, Kiev
  - Site Reference ID/Investigator# 30098, Kiev
  - Site Reference ID/Investigator# 30100, Kiev
  - Site Reference ID/Investigator# 30614, Kiev
  - Site Reference ID/Investigator# 30615, Kiev
  - Site Reference ID/Investigator# 30101, Kiev
  - Site Reference ID/Investigator# 22142, Kiev
  - Site Reference ID/Investigator# 30553, Kiev
  - Site Reference ID/Investigator# 30554, Kiev
  - Site Reference ID/Investigator# 30555, Kiev
  - Site Reference ID/Investigator# 30556, Kiev
  - Site Reference ID/Investigator# 30557, Kiev
  - Site Reference ID/Investigator# 30558, Kiev
  - Site Reference ID/Investigator# 30061, Kiev
  - Site Reference ID/Investigator# 30533, Kiev
  - Site Reference ID/Investigator# 30534, Kiev
  - Site Reference ID/Investigator# 30591, Kiev
  - Site Reference ID/Investigator# 30592, Kiev
  - Site Reference ID/Investigator# 30593, Kiev
  - Site Reference ID/Investigator# 30069, Kiev
  - Site Reference ID/Investigator# 30537, Kiev
  - Site Reference ID/Investigator# 30538, Kiev
  - Site Reference ID/Investigator# 30539, Kiev
  - Site Reference ID/Investigator# 30540, Kiev
  - Site Reference ID/Investigator# 29839, Kiev
  - Site Reference ID/Investigator# 30531, Kremenchuk
  - Site Reference ID/Investigator# 30532, Kremenchuk
  - Site Reference ID/Investigator# 40759, Kyiv
  - Site Reference ID/Investigator# 40760, Kyiv
  - Site Reference ID/Investigator# 30604, Luhansk
  - Site Reference ID/Investigator# 30605, Luhansk
  - Site Reference ID/Investigator# 30606, Luhansk
  - Site Reference ID/Investigator# 30559, Lviv
  - Site Reference ID/Investigator# 30561, Lviv
  - Site Reference ID/Investigator# 30562, Lviv
  - Site Reference ID/Investigator# 30563, Lviv
  - Site Reference ID/Investigator# 30564, Lviv
  - Site Reference ID/Investigator# 29948, Odesa
  - Site Reference ID/Investigator# 30055, Odesa
  - Site Reference ID/Investigator# 30062, Odesa
  - Site Reference ID/Investigator# 30594, Odesa
  - Site Reference ID/Investigator# 30595, Odesa
  - Site Reference ID/Investigator# 29838, Poltava
  - Site Reference ID/Investigator# 30044, Poltava
  - Site Reference ID/Investigator# 30045, Poltava
  - Site Reference ID/Investigator# 30063, Poltava
  - Site Reference ID/Investigator# 30126, Poltava
  - Site Reference ID/Investigator# 30618, Poltava
  - Site Reference ID/Investigator# 30619, Poltava
  - Site Reference ID/Investigator# 30620, Poltava
  - Site Reference ID/Investigator# 30621, Poltava
  - Site Reference ID/Investigator# 30072, Simferopol
  - Site Reference ID/Investigator# 30629, Vynnytsya
  - Site Reference ID/Investigator# 30631, Vynnytsya
  - Site Reference ID/Investigator# 30190, Yevpatoria
  - Site Reference ID/Investigator# 30068, Zaporizhya
  - Site Reference ID/Investigator# 30565, Zaporizhya
  - Site Reference ID/Investigator# 30566, Zaporizhya
  - Site Reference ID/Investigator# 30567, Zaporizhya
  - Site Reference ID/Investigator# 30568, Zaporizhya
  - Site Reference ID/Investigator# 30570, Zaporizhya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 2822 participants enrolled, 22 were excluded from analysis for the following reasons: No baseline data (11), did not meet inclusion criteria (7), missing or inconsistent inclusion/final data (2), and no Klacid SR treatment (2). The per-protocol population consists of 2800 participants.
Groups:
- Klacid SR: Participants with acute tracheitis, bronchitis, or pneumonia treated with Klacid SR
Period: Overall Study
Arm/Group | Klacid SR
Started | 2822
Completed | 2819
Not Completed | 3
Not completed — Did not take Klacid SR | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Klacid SR: The per-protocol population (2800 participants) with acute tracheitis, bronchitis, or pneumonia treated with Klacid SR.
Arm/Group | Klacid SR
Number analyzed (Participants) | 2800
Age Continuous [Mean (Standard Deviation); unit: years] — Based on the per-protocol population (2800 participants).
  years | 43.41 (13.79)
Age, Customized [Number; unit: Participants] — Based on the per-protocol population (2800 participants).
  Participants
    18 to 20 years | 64
    21 to 34 years | 763
    35 to 64 years | 1777
    65 to 84 years | 190
    85 years or older | 6
Sex/Gender, Customized [Number; unit: Participants] — The gender of the participants was not collected in this study.
  Participants
    Not reported | 2800
Region of Enrollment [Number; unit: Participants] — Based on the per-protocol population (2800 participants).
  Participants
    Ukraine | 2800

OUTCOME MEASURES:

1. Primary Outcome: Body Temperature
Description: Body temperature was measured at Visit 1 (initial visit) and at Visit 2 (approximately 10 to 16 days later, or as defined by the treating physician). Fever was defined as body temperature greater than or equal to 37 degrees Celsius/98.6 Fahrenheit. The presence or absence of fever is reported at Visit 1 and 2 for all participants and by age subgroups.
Time Frame: Visit 1 (initial visit), Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed. Visit 2 results are shown for those who had fever at Visit 1.
Measure: Number; unit: Participants
Groups:
- Klacid SR (Total): All participants with acute tracheitis, bronchitis, or pneumonia treated with Klacid SR.
- Klacid SR (18 to 64 Years of Age): Participants 18 to 64 years of age.
- Klacid SR (65 Years of Age or Older): Participants 65 years of age or older.
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Visit 1: No fever | 183 | 170 | 13
  Visit 1: Fever present | 2617 | 2434 | 183
  a) Fever resolved at Visit 2 | 1780 | 1655 | 125
  b) Fever still present at Visit 2 | 837 | 779 | 58

2. Primary Outcome: Cough and Its Character
Description: Participants were evaluated at Visit 1 (initial visit) and Visit 2 (10 to 16 days later or as defined by the treating physician). The presence of cough and the type of cough (productive, irritating, or both) was determined based on the clinical judgment of the treating physician. The presence or absence of cough are reported at Visits 1 and 2 for all participants and by age subgroups. For those participants who had a cough at Visit 1, the number of participants whose original type of cough subsequently resolved at Visit 2 is also presented.
Time Frame: Visit 1 (initial visit), Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Visit 1: Did not have cough | 118 | 110 | 8
  Visit 2: Did not have cough | 1813 | 1702 | 111
  Visit 1: Had irritating cough | 1671 | 1563 | 108
  Visit 2: Had irritating cough | 237 | 220 | 17
  Visit 1: Had productive cough | 1011 | 931 | 80
  Visit 2: Had productive cough | 749 | 682 | 67
  Visit 1: Had both types of cough | 0 | 0 | 0
  Visit 2: Had both types of cough | 1 | 0 | 1
  Had any cough at Visit 1 and resolved at Visit 2 | 1712 | 1609 | 103
  a) Irritating cough resolved at Visit 2 | 1438 | 1348 | 90
  b) Productive cough resolved at Visit 2 | 274 | 261 | 13

3. Primary Outcome: Dyspnoea
Description: Participants were evaluated at Visit 1 (initial visit) and Visit 2 (10 to 16 days later or as defined by the treating physician). The presence or absence of dyspnoea (difficulty breathing) was determined based on the clinical judgment of the treating physician and is reported for all participants and by age subgroup at Visit 1 and Visit 2. For participants with dyspnoea at Visit 1, whether the dyspnoea occurred at rest, after exercise, or both are reported. For those with dyspnoea at Visit 1, the number of participants whose original type of dyspnoea subsequently resolved at Visit 2 is noted.
Time Frame: Visit 1 (initial visit), Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Visit 1: No dyspnoea | 1821 | 1753 | 68
  Visit 2: No dyspnoea | 2608 | 2451 | 157
  Visit 1: Dyspnoea after exercise | 883 | 766 | 117
  Visit 2: Dyspnoea after exercise | 181 | 143 | 38
  Visit 1: Dyspnoea at rest | 95 | 85 | 10
  Visit 2: Dyspnoea at rest | 1 | 1 | 0
  Visit 1: Both types of dyspnoea | 1 | 0 | 1
  Visit 2: Both types of dyspnoea | 10 | 9 | 1
  Dyspnoea resolved at Visit 2 (either type) | 799 | 710 | 89
  a) After exercise dyspnoea resolved at Visit 2 | 705 | 626 | 79
  b) Resting dyspnoea resolved at Visit 2 | 94 | 84 | 10

4. Primary Outcome: Auscultation Findings
Description: Participants were evaluated at Visit 1 (initial visit) and Visit 2 (10 to 16 days later or as defined by the treating physician). The presence of abnormal breathing sounds such as wheezing or crackles was determined by the treating physician using auscultation (listening for sounds within the body, usually with a stethoscope in the chest, neck, or abdomen) combined with their clinical judgment. Results are reported at Visit 1 and Visit 2 for all participants and by age subgroups. For participants with abnormal breathing sounds at Visit 1, resolution was noted at Visit 2.
Time Frame: Visit 1 (initial visit), Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Visit 1: Normal breath sounds | 389 | 378 | 11
  Visit 2: Normal breath sounds | 2494 | 2350 | 144
  Visit 1: Wheezing | 1632 | 1518 | 114
  Visit 2: Wheezing | 184 | 153 | 31
  Visit 1: Crackles | 779 | 708 | 71
  Visit 2: Crackles | 122 | 101 | 21
  Abnormal breath sounds resolved at Visit 2 | 2108 | 1974 | 134
  a) Wheezing resolved at Visit 2 | 1449 | 1366 | 83
  b) Crackles resolved at Visit 2 | 659 | 608 | 51

5. Primary Outcome: Chest Xray - Necessary for Verification of the Diagnosis of Pneumonia , Community-acquired Pneumonia
Description: Chest xrays were taken at Visit 1 to determine the presence of absence of community-acquired pneumonia. Findings are presented for all participants and by age subgroups.
Time Frame: Visit 1 (Initial visit)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Findings did not indicate pneumonia | 1742 | 1651 | 91
  Findings indicated pneumonia | 1058 | 953 | 105

6. Primary Outcome: Previous Prescription of Other Antibiotic (Answer Whether Klacid SR is Given as the First or as Second Antibiotic)
Description: Treating physicians were asked if Klacid SR was the first or second antibiotic prescribed to treat the participant. Results are presented for all participants and age subgroups.
Time Frame: Visit 1 (Initial visit)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Klacid SR given as first antibiotic | 2381 | 2237 | 144
  Klacid SR given as second antibiotic | 377 | 327 | 50
  Klacid SR given as third antibiotic | 42 | 40 | 2

7. Primary Outcome: Therapeutic Response
Description: Therapeutic response (yes or no) was determined by the treating physician at Visit 2 based on the disappearance or significant alleviation of symptoms and regression of chest xray findings. The data are summarized by total number of participants and by age subgroups.
Time Frame: Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total) | Klacid SR (18 to 64 Years of Age) | Klacid SR (65 Years of Age or Older)
Number analyzed (Participants) | 2800 | 2604 | 196
Participants
  Had therapeutic response to therapy | 2786 | 2592 | 194
  No therapeutic response to therapy | 14 | 12 | 2

8. Secondary Outcome: Adverse Effects
Description: The number of participants experiencing adverse events, including serious adverse events, adverse events leading to study discontinuation, or adverse events leading to a dose reduction/temporarily stopping medication are summarized. See Reported Adverse Events for additional details.
Time Frame: Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total)
Number analyzed (Participants) | 2800
Participants
  Non-serious adverse events (AEs) | 14
  Serious AEs | 0
  Discontinued due to AEs | 1
  Dose reduced or stopped temporarily due to AEs | 0

9. Secondary Outcome: Compliance (Was the Dosage and Duration of Therapy Followed or Not; if Not - Explain the Reason)
Description: Compliance was assessed by asking physicians if participants took their medication as directed. If participants did not take their medication as directed, physicians were asked to give the reason.
Time Frame: Visit 2 (10th-16th day or any other day after Inclusion Visit defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total)
Number analyzed (Participants) | 2800
Participants
  Dosage was followed | 2786
  Dosage was not followed | 14
  a) Dosage not followed due to adverse event | 1
  b) Reason not reported | 13

10. Secondary Outcome: Termination of Treatment
Description: The number of participants who discontinued treatment is summarized.
Time Frame: Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Population: The per-protocol population was analyzed.
Measure: Number; unit: Participants
Arm/Group | Klacid SR (Total)
Number analyzed (Participants) | 2800
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected through Visit 2 (10th-16th day or any other day after Visit 1 defined by physician)
Description: The safety analysis set was used for the analysis of safety and tolerability. The safety population consisted of all subjects who received at least one dose of Klacid SR and had final visit documentation (2800 participants).
Arm/Group | Klacid SR
Serious Adverse Events (participants affected / at risk) | 0/2800
Other Adverse Events (participants affected / at risk) | 14/2800
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Klacid SR (N=2800)
Nausea (Gastrointestinal disorders) | 7
Dysgeusia (Nervous system disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 3
Disbacteriosis (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection